CLINICAL TRIAL: NCT00684983
Title: Randomized Phase II Trial of Capecitabine and Lapatinib With or Without IMC-A12 in Patients With HER2 Positive Breast Cancer Previously Treated With Trastuzumab and an Anthracycline and/or a Taxane
Brief Title: Capecitabine and Lapatinib Ditosylate With or Without Cixutumumab in Treating Patients With Previously Treated HER2-Positive Stage IIIB-IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00665; NCI-2009-00665 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PN0733_A15PAMDREVW01; NCCTG N0733; CDR0000596070; NCCTG-N0733; N0733 (Other: Alliance for Clinical Trials in Oncology); N0733 (Other: CTEP); U10CA180821 (NIH); U10CA025224 (NIH)
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: HER2 Positive Breast Carcinoma; Recurrent Breast Carcinoma; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
Keywords: IGF-1R; IMC-A12
MeSH Terms: conditions — Breast Neoplasms; Insulin-Like Growth Factor I, Resistance To | interventions — Capecitabine; cixutumumab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (lapatinib ditosylate, capecitabine) (Active Comparator): Patients receive capecitabine PO BID on days 1-14 and lapatinib ditosylate PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Lapatinib Ditosylate; Other: Quality-of-Life Assessment
- Arm B (cixutumumab, lapatinib ditosylate, capecitabine) (Experimental): Patients receive capecitabine and lapatinib ditosylate as in Arm A. Patients also receive cixutumumab IV over 1 hour on days 1, 8, and 15. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Biological: Cixutumumab; Drug: Lapatinib Ditosylate; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
  Arms: Arm B (cixutumumab, lapatinib ditosylate, capecitabine)
Drug: Lapatinib Ditosylate — Given PO
  Other Names: Tykerb
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies capecitabine and lapatinib ditosylate to see how well they work compared with capecitabine, lapatinib ditosylate, and cixutumumab in treating patients with previously treated HER2-positive stage IIIB-IV breast cancer. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with cixutumumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether capecitabine and lapatinib ditosylate are more effective when given with or without cixutumumab in treating breast cancer that has spread nearby or to other areas of the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression-free survival of HER2+ breast cancer patients randomized to receive lapatinib ditosylate (lapatinib) and capecitabine +/- cixutumumab (IMC-A12).

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of lapatinib and capecitabine +/- IMC-A12 in HER2+ breast cancer patients.

II. To compare the overall survival time, time to treatment failure, confirmed tumor response rate, and duration of response of lapatinib and capecitabine +/- IMC-A12 in HER2+ breast cancer patients.

III. To assess patient compliance per treatment arm and to compare overall quality of life and treatment side effects via patient-reported outcomes between treatment arms.

TRANSLATIONAL RESEARCH OBJECTIVES:

I. To determine the role of the following in predicting response to lapatinib and capecitabine +/- IMC-A12:

Ia. Expression patterns and/or activation IGF- and ErbB family of receptors and signaling molecules in formalin-fixed, paraffin-embedded breast tumor tissue.

Ib. Expression patterns and/or activation IGF- and ErbB receptors and signaling molecules in circulating tumor cells from breast cancer patients.

Ic. Changes in expression patterns and/or activation IGF- and ErbB receptors and signaling molecules following treatment with lapatinib and capecitabine +/- IMC-A12 in circulating tumor cells from breast cancer patients.

Id. Expression patterns of IGF-1, IGF-II, insulin, growth hormone, and the IGF binding proteins in the serum of breast cancer patients.

Ie. Changes in expression patterns of IGF-1, IGF-II, insulin, growth hormone, and the IGF binding proteins in the serum of breast cancer patients.

II. Banking of paraffin-embedded tissue blocks/slides and blood products (i.e., serum, plasma, and buffy coat) for future studies.

III. To assess the proportion of patients whose pathologic specimens were correctly diagnosed as HER2 positive (according to 2007 American Society of Clinical Oncology [ASCO] College of American Pathologist [CAP] guidelines) metastatic breast cancer.

OUTLINE: The first 10 patients enrolled on this study are assigned to cohort I (safety analysis). All other patients are assigned to cohort II (randomized treatment).

COHORT I (SAFETY ANALYSIS, closed to accrual): Patients receive cixutumumab intravenously (IV) over 1 hour on days 1, 8, and 15. Patients also receive capecitabine orally (PO) twice daily (BID) on days 1-14 and lapatinib ditosylate PO once daily (QD) on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

COHORT II (RANDOMIZED TREATMENT): Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive capecitabine PO BID on days 1-14 and lapatinib ditosylate PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive capecitabine and lapatinib ditosylate as in Arm A. Patients also receive cixutumumab IV over 1 hour on days 1, 8, and 15. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months until disease progression and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally advanced: (a T4 primary tumor and stage IIIB or IIIC disease) or metastatic breast cancer that has progressed after treatment with regimens that included trastuzumab and either an anthracycline or a taxane or both

  * NOTE: Agents need not have been given concurrently, nor in the same regimen
  * NOTE: Prior treatment with trastuzumab is required unless there is a contraindication for trastuzumab treatment
* Pre-treatment requirements:

  * Prior treatment with trastuzumab in the neo-adjuvant, adjuvant or metastatic setting is required

    * NOTE: Prior treatment with trastuzumab is required unless there is a contraindication for trastuzumab treatment
    * NOTE: Concomitant use of trastuzumab is not allowed in this study
  * Prior chemotherapy allowed in the neo-adjuvant, adjuvant, or metastatic setting; unlimited prior chemotherapy is allowed
  * Prior hormonal therapy allowed in the neo-adjuvant, adjuvant, or metastatic setting; unlimited prior hormonal therapy is allowed
  * HER2 positive, defined as:

    * Validated immunohistochemistry (IHC) assay score of 3+ (defined as uniform, intense staining of > 30% of invasive tumor cells)
    * -OR- Average HER2 gene copy number of > 6
    * -OR- Gene amplified (HER2:D17Z1 ratio > 2.20)
* Must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Hemoglobin > 9.0 g/dL (obtained =< 7 days prior to registration)
* White blood cells (WBC) >= 3,000/mL (obtained =< 7 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mL (obtained =< 7 days prior to registration)
* Platelet count >= 75,000/mL (obtained =< 7 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 7 days prior to registration)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x ULN or SGOT (AST) and SGPT (ALT) =< 5 x ULN if elevations are due to liver metastases (obtained =< 7 days prior to registration)
* Serum creatinine =< 1.5 x ULN (obtained =< 7 days prior to registration)
* Creatinine clearance >= 30 mL/min (calculated according to Cockcroft and Gault) (obtained =< 7 days prior to registration)

  * NOTE: In patients with moderate renal impairment (calculated creatinine clearance 30-50 mL/min) at baseline, a dose reduction of the capecitabine starting dose is required
* Fasting glucose < 120 mg/dL (obtained =< 7 days prior to registration)

  * NOTE: Patients with diabetes are allowed to participate, provided that their blood glucose is within the guidelines above upon enrollment
* International normalization ratio (INR) =< 1.5 x ULN (obtained =< 7 days prior to registration)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2
* Adequate cardiac function defined as an ejection fraction >= 50% as determined by multi gated acquisition scan (MUGA) or echocardiogram
* Life expectancy > 3 months
* Has written informed consent been obtained?
* Willingness to return to a North Central Cancer Treatment Group (NCCTG) or other participating cooperative group institution for treatment and follow-up
* Patient willing to provide tissue and blood samples for research purposes
* Availability of diagnostic material (i.e., diagnostic slides confirming locally advanced/metastatic disease and HER2 stained slides) and operative and pathology reports from diagnosis of locally advanced or metastatic breast cancer

  * NOTE: Biopsy of recurrent disease and submission of these materials is not required if materials available from initial diagnosis of locally advanced/metastatic disease
* Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (as determined by the treating physician)
* Stage III or IV invasive cancer, other than breast cancer, in =< 5 years prior to registration
* Actively being treated for other malignancy, excepting non-melanotic skin cancer or carcinoma-in-situ of the cervix; if there is a history of prior malignancy, patient must not be receiving other specific treatment for their cancer
* New York Heart Association class III or IV cardiovascular disease
* Current, active hepatic or biliary disease except Gilbert's syndrome or asymptomatic gallstones
* Evidence of active brain metastasis including leptomeningeal involvement; central nervous system (CNS) metastasis controlled by prior surgery and/or radiotherapy is allowed

  * NOTE: To be considered controlled, there must be at least 2 months of no symptoms or evidence of progression prior to study entry and corticosteroid therapy must have been discontinued
* Major surgery, chemotherapy, or immunologic therapy =< 4 weeks prior to registration
* Radiotherapy =< 4 weeks prior to registration, except if to a non-target lesion only; prior radiation to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed; if patient receives single dose radiation for palliation or radiation to non-target lesion, they may immediately proceed to registration without waiting; acute adverse events from radiation must have resolved to =< Common Terminology Criteria for Adverse Events (CTCAE) version (v) 3.0 grade 1
* Prior treatment with any therapy targeting IGF-I, IGF-II or its receptors (either monoclonal antibody or tyrosine kinase inhibitor), including but not limited to any of the following (which would have been received on a previous clinical trial):

  * IMC-A12 (cixutumumab)
  * CP-751,871 (figitumumab)
  * AMG-479
  * INSM-18
  * MK0646 (h7C10)
  * SCH717454 (19D12, robatumumab)
  * R1507
  * OSI-906
  * BMS-754807
  * PPP
  * NVP-AEW541
  * AVE-1642
  * MEDI-573
* Prior therapy with any therapy targeting HER1 (EGFR) and/or HER2 (either monoclonal antibody or tyrosine kinase) other than trastuzumab, including but not limited to any of the following:

  * Lapatinib (Tykerb)
  * Gefitinib (Iressa)
  * Erlotinib (Tarceva)
  * Cetuximab (Erbitux)
  * Panitumumab (Vectibix)
* Currently receiving treatment with any agents that are contraindicated by study therapies:

  * IMC-A12 - none identified to date
  * Lapatinib - CYP3A4 inhibitors and inducers, including grapefruit and grapefruit juice
  * Capecitabine - warfarin (Coumadin), cimetidine (Tagamet), allopurinol (Lopurin), sorivudine (Usevir) or brivudine (Brivex), ketoconazole (Nizoral), itraconazole (Sporanox), ritonavir (Norvir), amprenavir (Agenerase) or indinavir (Crixivan)
* Uncontrolled intercurrent illness including, but not limited to:

  * Poorly controlled diabetes
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of the safety of the prescribed regimens
* Currently receiving treatment in a different clinical study in which investigational procedures are performed or investigational therapies are administered
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive with an acquired immune deficiency syndrome (AIDS)-defining illness; HIV positive patients with cluster of differentiation (CD) 4 count within institutional normal range and no history of an AIDS-defining illness are eligible; however, some antiviral/antiretroviral medications which have CYP3A4 interactions are prohibited on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-07-30 (Actual); Primary Completion 2014-01-07 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tufia C Haddad, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (390):
- United States (390):
  - Providence Hospital, Mobile, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Salinas Valley Memorial, Salinas, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Lynn Regional Cancer Center - West, Boca Raton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Finley Hospital, Dubuque, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Cancer Trials Support Unit, Rockville, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Virtua Memorial, Mount Holly, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Staten Island University Hospital, Staten Island, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - McLeod Regional Medical Center, Florence, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford NCI Community Oncology Research Program of the North Central Plains, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Cancer Care-Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Haddad TC, He J, O'Sullivan CC, Chen B, Northfelt D, Dueck AC, Ballman KV, Tenner KS, Linden H, Sparano JA, Hopkins JO, De Silva C, Perez EA, Haluska P, Goetz MP. Randomized Phase II Trial of Capecitabine and Lapatinib with or without IMC-A12 (Cituxumumab) in Patients with HER2-Positive Advanced Breast Cancer Previously Treated with Trastuzumab and Chemotherapy: NCCTG N0733 (Alliance). Breast Cancer Res Treat. 2021 Jul;188(2):477-487. doi: 10.1007/s10549-021-06221-8. Epub 2021 Apr 14. PMID 33852121

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 68 (Arm A:20, B: 48) patients were accrued, 8 safety cohort patients from arm B are not eligible for primary end point analysis. There were 3 cancels (Arm B), 1 ineligible (arm A) and 1 major violation (Arm B, this patient is included in the primary analysis per protocol). Total of 64 patients started and completed the treatment.
Groups:
- Arm A: Patients receive oral capecitabine twice daily on days 1-14 and oral lapatinib ditosylate once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. lapatinib ditosylate: Given PO and capecitabine: Given PO
- Arm B: Patients receive capecitabine and lapatinib ditosylate as in arm I. Patients also receive cixutumumab IV over 1-1½ hours on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. cixutumumab: Given IV, lapatinib ditosylate: Given PO and capecitabine: Given PO
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 19 | 45
Completed | 19 | 45 (One major violation patient in Arm B is included in the primary analysis per protocol.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total of 68 patient were accrued. Three are cancels and one is ineligible. Sixty four (64) started the study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 19 | 45 | 64
Age, Continuous [Mean (Full Range); unit: years] | 57 [35 to 75] | 53 [29 to 78] | 53.5 [29 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 45 | 64
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 45 | 64

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Analysis of the primary endpoint, PFS, will be performed using Cox regression with treatment group as a single covariate.
Time Frame: From randomization to the earliest date of documentation of disease progression, up to 5 years
Population: First 8 patients in Arm B are from safety cohort, they are not eligible for primary end point
Measure: Median (95% Confidence Interval); unit: Median survival and CI in months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 19 | 37
Median survival and CI in months | 6.0 [4.3 to 8.6] | 4.9 [2.9 to 8.5]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Analysis of the primary endpoint, PFS, will be performed using Cox regression with treatment group as a single covariate; Test type: Superiority or Other; p = .89, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.58 to 1.89]

2. Secondary Outcome: Overall Survival
Description: Median Survival time (months)
Time Frame: From randomization to death due to any cause, up to 5 years
Population: All evaluable patients
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 19 | 37
Months | 16.8 [1.7 to 37.9] | 14.7 [3.1 to 47.7]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; p = 0.93, Log Rank; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.5 to 3]

3. Secondary Outcome: Time to Treatment Failure
Description: Distribution estimated by the Kaplan-Meier (1958) method for each treatment arm.
Time Frame: From the date of randomization to the date at which the patient is removed from treatment due to progression, adverse events, or refusal, up to 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 19 | 37
Months | 4.6 [0.4 to 12] | 4.4 [.8 to 24]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; p = .66, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [.53 to 1.92]

4. Secondary Outcome: Confirmed Tumor Response, Defined as Either a Complete Response (CR) or Partial Response (PR) Noted as the Objective Status on 2 Consecutive Evaluations at Least 6 Weeks Apart, Assessed by Response Evaluation Criteria for Solid Tumors (RECIST)
Time Frame: Up to 5 years
Population: Includes patients with at least one disease assessment at least 6 weeks after registration.
Measure: Number (95% Confidence Interval); unit: % of evaluable participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 16 | 31
% of evaluable participants | 43.8 [19.8 to 70.1] | 29 [14.2 to 48]

5. Secondary Outcome: Duration of Response
Description: Distribution estimated by the Kaplan-Meier (1958) method for each treatment arm.
Time Frame: Up to 5 years
Population: Evaluable patients that had a response to treatment drug
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 7 | 9
Months | 4.8 [3.2 to 8.6] | 6.9 [3 to 21.8]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Superiority; p = .26, Log Rank; Hazard Ratio (HR) = .39, 95% CI 2-sided [.09 to 1.53]

6. Secondary Outcome: Adverse Event Profile of Capecitabine and Lapatinib With and Without IMC-A12 (Using NCI CTCAE v3.0)
Description: All eligible patients that have initiated treatment will be considered evaluable for assessing adverse event rate(s) according to CTCAE v3.0 within each treatment arm. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
  4/19 (21.05%) 14/45 (31.11%)
Time Frame: Baseline to 30 days past end of treatment
Measure: Number; unit: percentage of patients with AEs
Groups:
- Arm I (Lapatinib Ditosylate, Capecitabine): Patients receive capecitabine PO BID on days 1-14 and lapatinib ditosylate PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Capecitabine: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Lapatinib Ditosylate: Given PO
  Quality-of-Life Assessment: Ancillary studies
- Arm II (Cixutumumab, Lapatinib Ditosylate, Capecitabine): Patients receive capecitabine and lapatinib ditosylate as in Arm I. Patients also receive cixutumumab IV over 1 hour on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Capecitabine: Given PO
  Cixutumumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Lapatinib Ditosylate: Given PO
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Arm I (Lapatinib Ditosylate, Capecitabine) | Arm II (Cixutumumab, Lapatinib Ditosylate, Capecitabine)
Number analyzed (Participants) | 19 | 45
percentage of patients with AEs | 21 | 31

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 4/19 | 14/45
Other Adverse Events (participants affected / at risk) | 19/19 | 43/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=19) | Arm B (N=45)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=19) | Arm B (N=45)
Hemoglobin decreased (Blood and lymphatic system disorders) | 11 (57) | 26 (137)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (3)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular bigeminy (Cardiac disorders) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 0 (0) | 2 (2)
Flashing vision (Eye disorders) | 0 (0) | 4 (12)
Vision blurred (Eye disorders) | 1 (2) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 8 (26)
Diarrhea (Gastrointestinal disorders) | 16 (46) | 35 (133)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (17)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (8)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 10 (20) | 21 (49)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 10 (14) | 22 (35)
Nausea (Gastrointestinal disorders) | 9 (11) | 22 (63)
Proctoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 9 (16)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (2) | 1 (1)
Fatigue (General disorders) | 17 (83) | 37 (175)
Fever (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 3 (5)
Pericardial pain (General disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (3)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 0 (0) | 1 (15)
Nail infection (Infections and infestations) | 0 (0) | 3 (12)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (8) | 10 (26)
Alkaline phosphatase increased (Investigations) | 0 (0) | 5 (7)
Amylase increased (Investigations) | 2 (3) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 9 (22) | 11 (21)
Bilirubin increased (Investigations) | 5 (12) | 6 (20)
Coagulopathy (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 5 (19)
INR increased (Investigations) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (6)
Leukocyte count decreased (Investigations) | 3 (3) | 6 (12)
Lipase increased (Investigations) | 2 (2) | 4 (4)
Lymphocyte count decreased (Investigations) | 1 (1) | 3 (7)
Neutrophil count decreased (Investigations) | 6 (19) | 9 (29)
Platelet count decreased (Investigations) | 2 (2) | 10 (31)
Serum cholesterol increased (Investigations) | 1 (1) | 3 (8)
Weight loss (Investigations) | 1 (1) | 11 (45)
Anorexia (Metabolism and nutrition disorders) | 2 (4) | 15 (46)
Blood glucose increased (Metabolism and nutrition disorders) | 9 (18) | 29 (131)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Glucose intolerance (Metabolism and nutrition disorders) | 2 (3) | 4 (21)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 4 (7)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 7 (10)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (2) | 5 (13)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (8)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 4 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (6)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (10)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (6) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (14) | 7 (13)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Taste alteration (Nervous system disorders) | 0 (0) | 11 (27)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (11)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (9)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (14)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (8)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (9)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (7) | 6 (11)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 14 (52) | 28 (118)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (28)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (7) | 9 (24)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (10)
Rash desquamating (Skin and subcutaneous tissue disorders) | 9 (20) | 21 (52)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (7)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (4)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less